CLINICAL TRIAL: NCT03384342
Title: Maintenance Therapy of Narrow-band UV-B Therapy in Patients With Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VC17DEDI0185
Record Dates: First submitted 2017-12-05; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Phototherapy; Vitiligo; Maintenance Therapy; Narrow-band UV-B
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): * For a total period of 12 months, perform Narrow-band UV-B therapy treatment once a month.
  * At this time, the dose of Narrow-band UV-B therapy therapy is based on the 50% of the maximum dose that the patient received for the treatment.
  Interventions: Device: Narrow-band UV-B therapy
- Control group (No Intervention): * Check for signs of enlarged vitiligo lesions at 3-month intervals for a total period of 12 months.
  * If recurrence of vitiligo is observed during the follow-up period, visit the clinic and check for recurrence.

INTERVENTIONS:
Device: Narrow-band UV-B therapy — * Patients treated with NBUVB and showed 75% or more repigmentation rate would be included.
  * For a total period of 12 months, narrow-band UV-B therapy is performed once a month.
  Arms: Experimental group

SUMMARY:
Although vitiligo is difficult to cure, recurrences are frequent after treatment, and many patients suffer from concerns about recurrence as well as disease. Psoriasis, another indication for ultraviolet radiation treatment, has been established that it can safely and effectively reduce the recurrence of psoriasis through monthly maintenance therapy.

The aim of this study was to evaluate the efficacy of Narrow-band UV-B therapy for the prevention of relapse in vitiligo.

DETAILED DESCRIPTION:
For a total period of 12 months, perform Narrow-band UV-B treatment once a month. Check for signs of enlarged vitiligo lesions at 3-month intervals for a total period of 12 months.

An independent evaluator will obtain the score of vitiligo area (Vitiligo Extent Score) from comparing clinical photographs of before registration and after the clinical trial, and judge whether vitiligo is recurred. This study is a randomized controlled trial, and the investigators plan to compare the recurrence rates of the experimental and control groups using the Chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age of 19 years or older
2. Patients of generalized vitiligo with lesions on the trunk
3. Patients who had treated with Narrow-band UV-B therapy previously and achieved more than 75% lesion improvement
4. Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

1. Patients under the age of 19
2. Patients with localized vitiligo and segmental vitiligo
3. Patients who are in a state of physical or mental impairment to perform treatment or pregnant
4. Patients with spreading of vitiligo lesions
5. Patients who do not want to do thie study or who refuse to write a consent form
6. Any other person deemed unsuitable for the examination at the discretion of the examiner

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-18 (Actual); Primary Completion 2018-11-18 (Estimated); Study Completion 2019-05-18 (Estimated)

PRIMARY OUTCOMES:
Recurrence of vitiligo | change from baseline area score at 12 months
  Clinical photographs taken before and 12 months after the completion of the study. The photographs will be used to measure the area of vitiligo lesion, and the investigators will compare the area score and judge whether or not there is a recurrence.

SECONDARY OUTCOMES:
The assessment of patient satisfaction | at baseline and at 12 months
  The assessment of patient satisfaction using five-point Likert scale. (Scale 1: strongly not-satisfied, Scale 2: Not-satisfied, Scale 3: Neither satisfied nor not-satisfied, Scale 4: Satisfied, Scale 5: Strongly satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Suwon, Gyonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No